CLINICAL TRIAL: NCT01417572
Title: Adjunctive Local Application of Lidocaine During Scleral Buckling Under General Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: isfahan university of medical sciences, isfahan university of medical sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 199
Record Dates: First submitted 2011-08-09; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2010-01

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- lidocaine (Experimental)
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: lidocaine — to evaluate the effect of lidocaine on oculocardiac reflex during the surgery

SUMMARY:
The purpose of this study is to evaluate the effect of topical lidocaine in scleral buckling surgery.

ELIGIBILITY:
Inclusion Criteria:

* Retinal detachment
* Retinal tear less than 3 hour clock

Exclusion Criteria:

* Vitreous hemorrhage
* Proliferative vitreoretinopathy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
intraoperative heart rate measurement | 6 month
decrease in pain and nausea,vomiting after surgery | 6 month
decrease in ocr after application of topical lidocaine | 6 month
postoperative nausea and vommitting | 6 month
postoperative pain | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran